CLINICAL TRIAL: NCT04072536
Title: Evaluation on Standardized Circuits of the Interest of a Robotic Module of Assistance to the Driving of Patients With Neurological Disorders, Regular Drivers of Electric Wheelchairs.
Brief Title: Evaluation on Standardized Circuits of the Interest of a Robotic Module of Assistance to the Driving
Acronym: SWADAPT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2019-A00476-51
Record Dates: First submitted 2019-06-21; First posted 2019-08-28 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Neurological Disorders
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Each patient included will test a wheelchair equipped with a collision avoidance assistance module in 2 conditions, assistance activated or not.
  This evaluation will be carried out in 3 standardized test circuits of increasing difficulty, one week apart. At each session, the patient will perform the circuit 6 times, including 3 with activated assistance, in a random order established upstream.
Who Masked: Participant, Outcomes Assessor
Masking Description: To minimize bias, this study will be randomized and conducted in single blind. The patient will not be aware of the activation or not of the assistance module placed on the electric wheelchair. Indeed, the investigative team will be in charge of the activation of the robotic module.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric wheelchair with activated assistance module (Experimental): This condition will be achieved in 3 standardized test circuits of increasing difficulty, one week apart. At each session, the patient will perform the circuit 6 times, including 3 with activated assistance, in a random order established upstream.
  Interventions: Device: Electric wheelchair with activated assistance module
- Electric wheelchair with assistance module not activated (Other): This condition will be achieved in 3 standardized test circuits of increasing difficulty, one week apart. At each session, the patient will perform the circuit 6 times, including 3 without activated assistance, in a random order established upstream.
  Interventions: Device: Electric wheelchair with assistance module not activated

INTERVENTIONS:
Device: Electric wheelchair with activated assistance module — This evaluation will be carried out in 3 standardized test circuits of increasing difficulty, one week apart. At each session, the patient will perform the circuit 6 times, including 3 with activated assistance
  Arms: Electric wheelchair with activated assistance module
Device: Electric wheelchair with assistance module not activated — This evaluation will be carried out in 3 standardized test circuits of increasing difficulty, one week apart. At each session, the patient will perform the circuit 6 times, including 3 with no activated assistance
  Arms: Electric wheelchair with assistance module not activated

SUMMARY:
The device that is the subject of this investigation is a robotic assistance module for driving a semi-autonomous electric wheelchair. This module is designed to accessorize the electric wheelchair to improve the safety conditions when driving an electric wheelchair, thus reducing the wheelchair accident rate on the one hand and facilitating access to the wheelchair to persons who can not claim it without the use of a safety device of this type.

DETAILED DESCRIPTION:
The device that is the subject of this investigation is a robotic assistance module for driving a semi-autonomous electric wheelchair. This module is designed to accessorize the electric wheelchair to improve the safety conditions when driving an electric wheelchair, thus reducing the wheelchair accident rate on the one hand and facilitating access to the wheelchair to persons who can not claim it without the use of a safety device of this type.

Each patient included will test a wheelchair equipped with a collision avoidance assistance module in 2 conditions, assistance activated or not. This evaluation will be carried out in 3 standardized test circuits of increasing difficulty, one week apart. At each session, the patient will perform the circuit 6 times, including 3 with activated assistance, in a random order established upstream.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18,
* Having freely consented to participate in the study,
* suffering from neurological disorders such as cerebro-lesion or neuro-degeneration,
* Having benefited from a prescription of electric wheelchair and circulating in an electric wheelchair for more than 3 months,
* of which the electric wheelchair is the main mode of transport,
* The physical measurements (weight, height) are compatible with the use of the electric wheelchair chosen for the development of the robotics assistance module.

Exclusion Criteria:

* Understanding difficulties preventing the realization of the protocol,
* Motor disorders of the upper limb requiring additional driving technical assistance,
* Patient having expressed difficulties impacting his safety of sedan and / or exterior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Number of collision | Day 1
  The primary judgment criterion is the number of collisions on different standardized circuits with and without activation of the robotic assistance module.
Number of collision | Day 8
  The primary judgment criterion is the number of collisions on different standardized circuits with and without activation of the robotic assistance module.
Number of collision | Day 15
  The primary judgment criterion is the number of collisions on different standardized circuits with and without activation of the robotic assistance module.

SECONDARY OUTCOMES:
Driving Speed | Day 1, Day 8 and Day 15
  Speed measured by the completion time of the course with and without activation of the assistance system on the different circuits
Wheelchair Skill Test | Day 1, Day 8 and Day 15
  Driving performance measured by the Wheelchair Skill Test items corresponding to the different courses, with and without activation of the assistance system
NASA-Task Load Index | Day 1, Day 8 and Day 15
  The cognitive load of tests under both conditions will be measured by the NASA-Task Load Index. It is in the form of six scales where the participant must assign a score between zero and one hundred to each of them, score indicating a growing level of intensity. Three dimensions relate to the demands imposed on the subject (mental, physical and temporal demands) and three to the interaction of a subject with the task (effort, frustration and performance)
Ease of Use Questionnaire | Day 1, Day 8 and Day 15
  The satisfaction of the use of the electric wheelchair under the conditions will be evaluated by the self-questionnaire Ease of Use Questionnaire. It measures the subjective usability of a product or service. It is a 30-item survey that examines four dimensions of usability: usefulness, ease of use, ease of learning, and satisfaction. The questionnaires were constructed as seven-point Likert rating scales. Users were asked to rate agreement with the statements, ranging from strongly disagree (1) to strongly agree (7).
UTAUT (Unified theory of acceptance of technology) questionnaire | Day 1, Day 8 and Day 15
  Questionnaire of acceptability / acceptance of the tool and its use by patients based on the Unified Theory of Acceptance and Use Technology (UTAUT).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pôle Saint-Hélier, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No